CLINICAL TRIAL: NCT04998357
Title: Study Title: Autologous Mitochondrial Transplant for Cerebral Ischemia
Brief Title: Autologous Mitochondrial Transplant for Cerebral Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Melanie Walker, Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006638
Record Dates: First submitted 2021-07-21; First posted 2021-08-10 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Ischemia
Keywords: autologous mitochondrial transplantation; ischemic stroke
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transplantation (Experimental): Endovascular infusion
  Interventions: Other: Endovascular autologous mitochondrial transplantation

INTERVENTIONS:
Other: Endovascular autologous mitochondrial transplantation — During standard-of-care endovascular reperfusion procedure, subjects will have autologous mitochondria infused via microcatheter into ischemic brain.

SUMMARY:
The investigators propose to infuse healthy autologous mitochondria into cerebral vessels supplying brain tissue experiencing ischemia in patients who undergo standard-of- care endovascular reperfusion therapy.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of morbidity and mortality worldwide. More than 80% of strokes are the result of ischemia caused by blockage of one or more cerebral arteries. Lack of blood supply starves brain cells of necessary glucose and oxygen, and disturbs cellular homeostasis, eventually resulting in neuronal death.

Mitochondria are tiny organelles present in nearly all types of human cells and are vital to our survival. Much like a battery, they generate most of our adenosine triphosphate (ATP), the energy currency of the cell. Mitochondria are also involved in other tasks, such as signaling between cells and cell death. All these functions can be impaired during ischemia because of the damage caused to mitochondria.

Based on many preclinical studies in animals, damage caused by ischemia can be reversed after infusing healthy mitochondria into injured tissues. An ongoing clinical trial in human hearts at Boston Children's Hospital has also demonstrated that transplanting autologous mitochondria via infusion or direct injection is well-tolerated and safe.

The investigators at the University of Washington are recruiting subjects for a first-in-human-brain trial to confirm the safety of autologous mitochondrial transplant during brain ischemia. The transplantation will be performed within the same procedure as the clinically indicated reperfusion treatment.

During standard-of-care endovascular treatment for cerebral ischemia, the investigators will obtain a very small biopsy from the muscle tissue adjacent to our surgical access site. Muscle tissue will be processed at bedside to extract the autologous mitochondria as performed in prior human cardiac trial and validated in animal studies. The endovascular treatment proceeds without disruption as clinically indicated, and the mitochondria are infused into the brain artery via micro-catheter during reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for endovascular thrombectomy to treat acute large vessel occlusion
* Eligible for angioplasty (microcatheter-based balloon/mechanical and chemical angioplasty) to treat acute cerebral vasospasm after aneurysmal subarachnoid hemorrhage
* Subjects for whom there is likely to be enough time to obtain meaningful consent from patient or legally-authorized representative

Exclusion Criteria:

* Unable to receive a brain MRI scan
* Known mitochondrial disease
* Hemodynamically unstable patients in whom standard of care endovascular reperfusion treatment cannot safely be performed or completed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe adverse events during mitochondrial infusion | Through completion of reperfusion therapy, up to one hour post-infusion
  Cerebral angiography is performed and reviewed in real-time throughout the standard of care reperfusion treatment, including before and after microcatheter infusion of mitochondria.
Incidence of severe adverse vascular events immediately post-mitochondrial infusion | Up to 3 hours post-mitochondrial infusion
  Post-reperfusion therapy, CT scans are performed as part of the standard of care. The post-procedure CT scan will be reviewed for severe adverse events associated with the microcatheter infusion of mitochondria.
Incidence of severe systemic adverse events associated with mitochondrial infusion | Up to seven days after procedure completion
  Post-reperfusion therapy, peripheral blood studies are performed and reviewed as part of the standard of care to assess systemic function. These include complete blood counts, coagulation studies, and serum chemistry.
Incidence of severe adverse events related to muscle biopsy | Up to six hours after procedure completion
  Muscle biopsy is obtained through the same incision as vascular access. The access site is evaluated via physical examination by medical personnel for six hours post-intervention per standard of care protocol.

SECONDARY OUTCOMES:
Reduction of infarct volume post-mitochondrial infusion | Up to seven days after procedure completion.
  Patients undergo brain MRI as part of standard of care evaluation after reperfusion therapy. These studies are compared with initial brain imaging studies obtained prior to reperfusion therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie S Walker, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miralles FJ, Prijoles KL, Winter A, Levitt MR, Sancak Y, Walker M. Periprocedural therapeutics do not impair extracellular mitochondrial viability in transplantation. J Cereb Blood Flow Metab. 2025 May 14:271678X251340232. doi: 10.1177/0271678X251340232. Online ahead of print. PMID 40367391
- [Background] Walker, M., Federico, E., Sancak, Y. et al. Mitochondrial Transplantation in Ischemic Stroke: Insights from a First-in-Human Brain Trial. Curr Transpl Rep 11, 53-62 (2024). https://doi.org/10.1007/s40472-024-00428-6
- [Background] Walker M, Levitt MR, Federico EM, Miralles FJ, Levy SH, Lynne Prijoles K, Winter A, Swicord JK, Sancak Y. Autologous mitochondrial transplant for acute cerebral ischemia: Phase 1 trial results and review. J Cereb Blood Flow Metab. 2024 Dec 4:271678X241305230. doi: 10.1177/0271678X241305230. Online ahead of print. PMID 39628322
- [Background] Preble JM, Pacak CA, Kondo H, MacKay AA, Cowan DB, McCully JD. Rapid isolation and purification of mitochondria for transplantation by tissue dissociation and differential filtration. J Vis Exp. 2014 Sep 6;(91):e51682. doi: 10.3791/51682. PMID 25225817
- [Background] Guariento A, Piekarski BL, Doulamis IP, Blitzer D, Ferraro AM, Harrild DM, Zurakowski D, Del Nido PJ, McCully JD, Emani SM. Autologous mitochondrial transplantation for cardiogenic shock in pediatric patients following ischemia-reperfusion injury. J Thorac Cardiovasc Surg. 2021 Sep;162(3):992-1001. doi: 10.1016/j.jtcvs.2020.10.151. Epub 2020 Dec 1. PMID 33349443
- [Background] Weixler V, Lapusca R, Grangl G, Guariento A, Saeed MY, Cowan DB, Del Nido PJ, McCully JD, Friehs I. Autogenous mitochondria transplantation for treatment of right heart failure. J Thorac Cardiovasc Surg. 2021 Jul;162(1):e111-e121. doi: 10.1016/j.jtcvs.2020.08.011. Epub 2020 Aug 10. PMID 32919774
- [Background] Doulamis IP, Guariento A, Duignan T, Kido T, Orfany A, Saeed MY, Weixler VH, Blitzer D, Shin B, Snay ER, Inkster JA, Packard AB, Zurakowski D, Rousselle T, Bajwa A, Parikh SM, Stillman IE, Del Nido PJ, McCully JD. Mitochondrial transplantation by intra-arterial injection for acute kidney injury. Am J Physiol Renal Physiol. 2020 Sep 1;319(3):F403-F413. doi: 10.1152/ajprenal.00255.2020. Epub 2020 Jul 20. PMID 32686525
- [Background] Orfany A, Arriola CG, Doulamis IP, Guariento A, Ramirez-Barbieri G, Moskowitzova K, Shin B, Blitzer D, Rogers C, Del Nido PJ, McCully JD. Mitochondrial transplantation ameliorates acute limb ischemia. J Vasc Surg. 2020 Mar;71(3):1014-1026. doi: 10.1016/j.jvs.2019.03.079. Epub 2019 Jul 26. PMID 31353269
- [Background] Ramirez-Barbieri G, Moskowitzova K, Shin B, Blitzer D, Orfany A, Guariento A, Iken K, Friehs I, Zurakowski D, Del Nido PJ, McCully JD. Alloreactivity and allorecognition of syngeneic and allogeneic mitochondria. Mitochondrion. 2019 May;46:103-115. doi: 10.1016/j.mito.2018.03.002. Epub 2018 Mar 26. PMID 29588218
- [Background] McCully JD, Levitsky S, Del Nido PJ, Cowan DB. Mitochondrial transplantation for therapeutic use. Clin Transl Med. 2016 Mar;5(1):16. doi: 10.1186/s40169-016-0095-4. Epub 2016 Apr 29. PMID 27130633
- [Background] Hayakawa K, Esposito E, Wang X, Terasaki Y, Liu Y, Xing C, Ji X, Lo EH. Transfer of mitochondria from astrocytes to neurons after stroke. Nature. 2016 Jul 28;535(7613):551-5. doi: 10.1038/nature18928. PMID 27466127
- [Background] Pluchino S, Peruzzotti-Jametti L, Frezza C. Astrocyte power fuels neurons during stroke. Swiss Med Wkly. 2016 Nov 10;146:w14374. doi: 10.4414/smw.2016.14374. eCollection 2016. No abstract available. PMID 27878792
- [Background] Bambrick L, Kristian T, Fiskum G. Astrocyte mitochondrial mechanisms of ischemic brain injury and neuroprotection. Neurochem Res. 2004 Mar;29(3):601-8. doi: 10.1023/b:nere.0000014830.06376.e6. PMID 15038607
- [Background] Wu M, Gu X, Ma Z. Mitochondrial Quality Control in Cerebral Ischemia-Reperfusion Injury. Mol Neurobiol. 2021 Oct;58(10):5253-5271. doi: 10.1007/s12035-021-02494-8. Epub 2021 Jul 18. PMID 34275087
- [Background] Norat P, Soldozy S, Sokolowski JD, Gorick CM, Kumar JS, Chae Y, Yagmurlu K, Prada F, Walker M, Levitt MR, Price RJ, Tvrdik P, Kalani MYS. Mitochondrial dysfunction in neurological disorders: Exploring mitochondrial transplantation. NPJ Regen Med. 2020 Nov 23;5(1):22. doi: 10.1038/s41536-020-00107-x. PMID 33298971
- [Background] Norat P, Sokolowski JD, Gorick CM, Soldozy S, Kumar JS, Chae Y, Yagmurlu K, Nilak J, Sharifi KA, Walker M, Levitt MR, Klibanov AL, Yan Z, Price RJ, Tvrdik P, Kalani MYS. Intraarterial Transplantation of Mitochondria After Ischemic Stroke Reduces Cerebral Infarction. Stroke Vasc Interv Neurol. 2023 May;3(3):e000644. doi: 10.1161/svin.122.000644. Epub 2023 Mar 2. PMID 37545759
- See also: The Stroke & Applied NeuroScience Center at the University of Washington — https://sanscenter.org/